CLINICAL TRIAL: NCT03158025
Title: A Randomized, Double-Blind, 6-Way Crossover Study to Determine the Abuse Potential of Single Oral Doses of Lemborexant Compared to Zolpidem, Suvorexant and Placebo in Healthy, Non-Dependent, Recreational Sedative Users
Brief Title: A Study to Determine the Abuse Potential of Single Oral Doses of Lemborexant Compared to Zolpidem, Suvorexant and Placebo in Healthy, Non-Dependent, Recreational Sedative Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2006-A001-103
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2018-07

CONDITIONS: Insomnia Disorders
Keywords: Recreational sedatives; Healthy participants; Lemborexant; E2006; Zolpidem; Suvorexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; suvorexant; lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo, LEM 10 mg, SUV 40 mg, LEM 20 mg, ZOL 30 mg, LEM 30 mg (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: Placebo (3 × placebo lemborexant [LEM] tablets; 3 × placebo zolpidem [ZOL] tablets; 2 × placebo suvorexant [SUV], over-encapsulated); LEM 10 milligrams (mg) (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets); LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated); LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant
- LEM 10 mg, LEM 20 mg, Placebo, LEM 30 mg, SUV 40 mg, ZOL 30 mg (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: LEM 10 mg (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); placebo (3 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets); ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant
- LEM 20 mg, LEM 30 mg, LEM 10 mg, ZOL 30 mg, Placebo, SUV 40 mg (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 10 mg (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated); placebo (3 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant
- LEM 30 mg, ZOL 30 mg, LEM 20 mg, SUV 40 mg, LEM 10 mg, Placebo (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated); LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets); LEM 10 mg (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); placebo (3 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant
- ZOL 30 mg, SUV 40 mg, LEM 30 mg, Placebo, LEM 20 mg, LEM 10 mg (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated); SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets); LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); placebo (3 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 10 mg (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant
- SUV 40 mg, Placebo, ZOL 30 mg, LEM 10 mg, LEM 30 mg, LEM 20 mg (Experimental): Participants will receive the following treatments (orally) in Treatments Periods 1 through 6, respectively: SUV 40 mg (2 × 20 mg SUV tablets, over-encapsulated; 3 × placebo ZOL tablets; 3 × placebo LEM tablets); placebo (3 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); ZOL 30 mg (3 × 10 mg ZOL tablets; 3 × placebo LEM tablets; 2 × placebo SUV, over-encapsulated); LEM 10 mg (1 × 10 mg LEM tablet; 2 × placebo LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 30 mg (3 × 10 mg LEM tablets; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated); LEM 20 mg (2 × 10 mg LEM tablets; 1 × placebo LEM tablet; 3 × placebo ZOL tablets; 2 × placebo SUV, over-encapsulated). Each treatment period will be separated by a washout interval of at least 14 days.
  Interventions: Drug: Zolpidem tablets; Drug: Suvorexant tablets, over-encapsulated; Drug: Lemborexant tablets; Drug: Placebo lemborexant; Drug: Placebo zolpidem; Drug: Placebo suvorexant

INTERVENTIONS:
Drug: Zolpidem tablets — Zolpidem 3 x 10 mg tablets will be administered orally.
  Other Names: AMBIEN; zolpidem tartrate
Drug: Suvorexant tablets, over-encapsulated — Suvorexant 2 x 20 mg tablets, over-encapsulated, will be administered orally.
  Other Names: BELSOMRA
Drug: Lemborexant tablets — Lemborexant 1 x 10 mg, 2 x 10 mg, or 3 x 10 mg tablets will be administered orally.
  Other Names: E2006
Drug: Placebo lemborexant — Placebo 1 x 10 mg, 2 x 10 mg, or 3 x 10 mg lemborexant tablets will be administered orally.
Drug: Placebo zolpidem — Placebo 3 x 10 mg zolpidem tablets will be administered orally.
Drug: Placebo suvorexant — Placebo 2 x 20 mg suvorexant tablets, over-encapsulated, will be administered orally.

SUMMARY:
The primary purpose of this study is to evaluate the abuse potential of lemborexant (E2006) in comparison to placebo and 2 controls with known abuse potential (ie, zolpidem and suvorexant) with similar indications (zolpidem and suvorexant) or mechanisms of action (suvorexant).

DETAILED DESCRIPTION:
This is a single-center, single oral dose, randomized, double-blind, placebo-controlled, 6-way crossover study in healthy, non-dependent recreational sedative users.

ELIGIBILITY:
Inclusion Criteria

* Healthy, male or female, 18 to 55 years of age, inclusive, at the time of informed consent
* Current sedative users who have used sedatives (e.g., zolpidem, benzodiazepines) for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least five times in the past year and used sedatives for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least once in the 12 weeks before Screening.
* A body mass index (BMI) of 18.0 to 33.0 kilograms per meters squared (kg/m^2), inclusive, and a minimum weight of 50.0 kg at Screening
* Female participants of childbearing potential with male sexual partners must be using and willing to continue using highly effective contraception for at least 1 month prior to Screening and for at least 1 month after the last study drug administration
* Female participants of non-childbearing potential must meet specified criteria.
* Male participants with female sexual partners of childbearing potential must be using and willing to continue using highly effective contraception from Screening and for at least 1 month after the last study drug administration.
* Participants who are using hormonal contraceptives must be on a stable dose of the same hormonal contraceptive product for at least 1 month before dosing and agree to use the same contraceptive during the study and for at least 1 month after the last study drug discontinuation
* Demonstrate the following in the Qualification Period:

  1. Ability to distinguish orally administered zolpidem 30 mg and suvorexant 40 mg from placebo on the bipolar Drug Liking (at this moment) Visual analog scale (VAS), defined as a ≥15 point peak increase for Drug Liking in response to zolpidem and suvorexant relative to placebo following drug administration. A peak score of ≥65 must be indicated on the bipolar measure of Drug Liking (at this moment) in response to zolpidem and suvorexant
  2. Display an acceptable placebo response, defined as a VAS response between 40 to 60 inclusive, for peak (Emax) Drug Liking (at this moment)
  3. Demonstrate responses to zolpidem and suvorexant that are consistent with discrimination relative to placebo on other subjective measures, as judged by the study center staff
  4. Tolerate study treatment (eg, no episodes of vomiting within the first 3 hours postdose) and demonstrate ability to complete the pharmacodynamic assessments (eg, no unarousable sedation within 4 hours postdose)
  5. Demonstrate general behavior suggestive that the participant could successfully complete the study, as judged by the study center staff.
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments
* Must provide written informed consent prior to the initiation of any protocol-specific procedures

Exclusion Criteria

* Substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition Text Revision (DSM IV-TR), and/or have ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence
* Female participants who are currently pregnant (have a positive pregnancy test) or lactating or who are planning to become pregnant within 1 month of the last study drug administration. No ovum donation is allowed during the study period and for 1 month after study drug discontinuation.
* Male participants who have not had a successful vasectomy (self-reported, confirmed azoospermia) or they and their female partners do not meet specified Inclusion Criteria (i.e., not practicing highly effective contraception throughout the study period and for 1 month after study drug discontinuation). No sperm donation is allowed during the study period and for 1 month after study drug discontinuation.
* Are currently abstinent and do not agree to use a highly effective form of contraception or refrain from sexual activity during the study period and for 1 month after study drug discontinuation
* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
* History of gastrointestinal surgery, or evidence of disease that may influence the outcome of the study, within 4 weeks before dosing (e.g., psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism)
* Participated in, is currently participating in, or is seeking treatment for substance- or alcohol-related disorders (excluding nicotine and caffeine)
* Heavy smokers (≥20 cigarettes or eCigarettes per day on average in the past 30 days before Screening), chews tobacco, uses a nicotine transdermal patch (including nicotine-containing products), or is unable to abstain from smoking for at least 8 hours during any day
* Participant is a habitual napper (i.e., habitually naps more than 3 times per week)

  a. Self-reported insomnia disorder, breathing-related sleep disorders, periodic limb movement disorder, restless legs syndrome, nightmare disorder, non-rapid eye movement (REM) sleep arousal disorders (sleep terror disorder or sleepwalking disorder), REM sleep behavior disorder, circadian rhythm sleep-wake disorders, or narcolepsy as defined by the DSM-Fifth Edition (DSM 5), or an exclusionary score (as detailed below) on any of the following subscales of the SLEEP50 Questionnaire:
  1. ≥15 on Apnea subscale
  2. ≥19 on Insomnia subscale if and only if also ≥15 on Impact subscale
  3. ≥7 on Narcolepsy subscale
  4. ≥7 on Restless Legs Syndrome (RLS) or Periodic Limb Movement Disorder (PLMD) subscale
  5. ≥8 on Circadian Rhythm subscale
  6. ≥7 on Sleepwalking subscale
  7. ≥3 on Item 32 and ≥9 on Items 33 to 35 (i.e., on nightmare subscale)
  8. ≥15 on Impact subscale
* Has been diagnosed with cancer within 3 years before Screening (excluding treated squamous or basal cell carcinoma of the skin), or has an active malignancy of any type (including squamous or basal cell carcinoma of the skin)
* Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding (i.e., QTcF >450 milliseconds [msec]), or laboratory test results that require medical treatment at Screening or that, in the opinion of the investigator, could affect the safety of the participant or the validity of the study
* Increased respiratory impairment risk, including those with sleep apnea or myasthenia gravis
* Participants with any history of suicidal ideation or suicidal behavior (lifetime and 12 months), as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS; Screening version)
* Known hypersensitivity or known allergy to zolpidem, suvorexant, or other sedative-hypnotics (eg, benzodiazepines) or study drug excipients (eg, lactose)
* Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Require concomitant treatment with moderate and strong cytochrome P450 (CYP) 3A4, 2C9, 2C19, 1A2, and 2D6 inhibitors or any inducer, or respiratory depressants, or cannot safely discontinue prohibited substances within the washout interval before receiving study drug, according to the Investigator or designee. Medications that may interact with study drugs include but are not limited to imipramine, chlorpromazine, sertraline, fluoxetine, rifampin, and ketoconazole. Use of prohibited medication within 30 days prior to screening; use of any other antihistamine, anticholinergic, melatonin, dehydroepiandrosterone (DHA), or herbal sleep or relaxation remedy within 7 days before screening will also be exclusionary at the discretion of the Investigator or designee.
* Received treatment with an investigational drug within 30 days, an investigational antibody treatment within 6 months, or 5-half-lives (if the half-life is known), whichever is longer, preceding the first dose of study
* Donated or had a loss of more than 500 milliliters (mL) of whole blood within 30 days before entry into the Treatment Phase
* Unwilling to be searched (including personal effects) for illicit substances before admission to the study center or during the participants' stay at the clinic
* In the opinion of the Principal Investigator (PI) or designee, are considered unsuitable or unlikely to comply with the study protocol for any reason, including compliance with the Study Restrictions and Prohibitions
* Do not abstain from alcohol for 24 hours before Screening as confirmed by a positive alcohol breath test (Note: Participants that do not meet this criterion may be re-screened at a later date).
* Difficulty with venous blood draws
* An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Do not agree to abstain from recreational drug use throughout the study, from Screening until after the last visit
* A participant who, in the opinion of the PI or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason
* Current pending legal charges or who are currently on probation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Mean peak Maximum Effect (Emax) score for Drug Liking on a Visual Analog Scale (VAS) | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis is conducted to evaluate abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."

SECONDARY OUTCOMES:
Mean time to peak effect (TEmax) score for Drug Liking on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."
Mean peak minimum effect (Emin) score for Drug Liking on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."
Mean time to peak minimum effect (TEmin) score for Drug Liking on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."
Mean time-averaged area under the effects curve (TA_AUE) score for Drug Liking on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."
Mean Emax score for Overall Drug Liking (Overall, my liking for this drug is) on a VAS | 12 (Day 1), 24 (Day 2), and 48 hours (Day 3) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "Overall, my liking for this drug is." The VAS will be scored as an integer from 0 (strong disliking) to 100 (strong liking). The neutral point equals 50 and will be labeled with the anchor "neither like nor dislike."
Mean Emax score for taking the drug again on a VAS | 12 (Day 1), 24 (Day 2), and 48 hours (Day 3) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "I would take this drug again." The VAS will be scored as an integer from 0 (definitely not) to 100 (definitely so). The neutral point equals 50 and will be labeled with the anchor "neutral."
Mean Emax score for Subjective Drug Value (SDV) | 12 (Day 1), 24 (Day 2), and 48 hours (Day 3) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to choose between theoretically receiving another dose of the drug to take home or an envelope containing a specified amount of money. Depending on the answer to each question, the monetary value in the next question will be either higher or lower.
Mean Emax score for Good Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel good drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TEmax score for Good Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel good drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TA_AUE score for Good Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel good drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean Emax score for Feeling Stoned on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel stoned." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TEmax score for Feeling Stoned on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel stoned." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TA_AUE score for Feeling Stoned on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel stoned." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean Emax score for Feeling High on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel high." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TEmax score for Feeling High on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel high." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TA_AUE score for Feeling High on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel high." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean Emax score for Bad Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel bad drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TEmax score for Bad Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel bad drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean TA_AUE score for Bad Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel bad drug effects." The VAS will be scored as an integer from 0 (not at all) to 100 (extremely).
Mean Emax score for Sedative Effect on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my mental state is…." The VAS will be scored as an integer from 0 (very drowsy) to 100 (very alert). The neutral point equals 50 and will be labeled with "Neither drowsy nor alert."
Mean TEmax score for Sedative Effect on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my mental state is…." The VAS will be scored as an integer from 0 (very drowsy) to 100 (very alert). The neutral point equals 50 and will be labeled with "Neither drowsy nor alert."
Mean TA_AUE score for Sedative Effect on a VAS | Pre-dose; 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, my mental state is…." The VAS will be scored as an integer from 0 (very drowsy) to 100 (very alert). The neutral point equals 50 and will be labeled with "Neither drowsy nor alert."
Mean Emax for Addiction Research Center Inventory (ARCI) Pentobarbital-Chlorpromazine-Alcohol Group (PCAG) subscale score | 1, 2, 4, and 8 hours (all Day 1) post-dose of each treatment cycle (up to 11 weeks)
  The shortened version of the ARCI contains the PCAG scale, consisting of 15 items measuring sedation effects. Participants indicate their responses by selecting "True" or "False" with a mouse. One point is given for each response that agrees with the scoring direction on the scale (i.e., True items receive a score of 1 if the answer is "True"; False items receive a score of 1 if the answer is "False"; no points are given when the answer is opposite to the scoring direction).
Mean TEmax for ARCI PCAG subscale score | 1, 2, 4, and 8 hours (all Day 1) post-dose of each treatment cycle (up to 11 weeks)
  The shortened version of the ARCI contains the PCAG scale, consisting of 15 items measuring sedation effects. Participants indicate their responses by selecting "True" or "False" with a mouse. One point is given for each response that agrees with the scoring direction on the scale (i.e., True items receive a score of 1 if the answer is "True"; False items receive a score of 1 if the answer is "False"; no points are given when the answer is opposite to the scoring direction).
Mean TA-AUE for ARCI PCAG subscale score | 1, 2, 4, and 8 hours (all Day 1) post-dose of each treatment cycle (up to 11 weeks)
  The shortened version of the ARCI contains the PCAG scale, consisting of 15 items measuring sedation effects. Participants indicate their responses by selecting "True" or "False" with a mouse. One point is given for each response that agrees with the scoring direction on the scale (i.e., True items receive a score of 1 if the answer is "True"; False items receive a score of 1 if the answer is "False"; no points are given when the answer is opposite to the scoring direction).
Mean Emax score for Any Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel any drug effect" The VAS will be scored as an integer from 0 (not at all) to 100 (extremely)
Mean TEmax score for Any Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel any drug effect" The VAS will be scored as an integer from 0 (not at all) to 100 (extremely)
Mean TA_AUE score for Any Effects on a VAS | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  Analysis will be conducted to evaluate objective and subjective effects related to abuse potential. Participants will be asked to respond to the following question on a VAS: "At this moment, I feel any drug effect" The VAS will be scored as an integer from 0 (not at all) to 100 (extremely)
Mean Emax score for Observer's Assessment of Alertness/Sedation (OAA/S): composite and sum scores | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The OAA/S Scale was developed to measure the level of alertness in participants who are sedated. The OAA/S scale is composed of the following assessment categories: responsiveness, speech, facial expression, and eyes. The OAA/S scale will be scored in 2 ways: a composite score (from 1 [less alert] to 5 [alert]), defined as the lowest score in any one of the 4 assessment categories; and a sum score, which is calculated as the total of the scores in the 4 assessment categories (from 4 [less alert] to 20 [more alert]).
Mean TA_AUE score for OAA/S: composite and sum scores | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The OAA/S Scale was developed to measure the level of alertness in participants who are sedated. The OAA/S scale is composed of the following assessment categories: responsiveness, speech, facial expression, and eyes. The OAA/S scale will be scored in 2 ways: a composite score (from 1 [less alert] to 5 [alert]), defined as the lowest score in any one of the 4 assessment categories; and a sum score, which is calculated as the total of the scores in the 4 assessment categories (from 4 [less alert] to 20 [more alert]).
Maximum change from baseline (CFBmax) in Choice Reaction Time (CRT) score (Motor Reaction Time [MRT] subscale score, Recognition Reaction Time [RRT] subscale score, and Total Reaction Time [TRT] subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The CRT task is a classic test of reaction time used to measure psychomotor performance. During this test, the participant is presented with an onscreen equivalent of the numeric keypad. The participant must quickly press the buttons on a separate keypad that corresponds with the keys illuminated on the screen. The CRT task comprises 3 outcome variables: RRT, MRT, and TRT. RRT is the time it takes for a participant to notice the light (i.e., the time between stimulus onset and the participant lifting his or her finger from the start button). MRT indexes the movement component of this task and is the time between the participant lifting his or her finger from the start button and touching the response button. TRT is the sum of RRT and MRT.
Mean TA_AUE of CRT score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The CRT task is a classic test of reaction time used to measure psychomotor performance. During this test, the participant is presented with an onscreen equivalent of the numeric keypad. The participant must quickly press the buttons on a separate keypad that corresponds with the keys illuminated on the screen. The CRT task comprises 3 outcome variables: RRT, MRT, and TRT. RRT is the time it takes for a participant to notice the light (i.e., the time between stimulus onset and the participant lifting his or her finger from the start button). MRT indexes the movement component of this task and is the time between the participant lifting his or her finger from the start button and touching the response button. TRT is the sum of RRT and MRT.
Minimum change from baseline (CFBmin) of percentage correct response relative to CRT score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The CRT task is a classic test of reaction time used to measure psychomotor performance. During this test, the participant is presented with an onscreen equivalent of the numeric keypad. The participant must quickly press the buttons on a separate keypad that corresponds with the keys illuminated on the screen. The CRT task comprises 3 outcome variables: RRT, MRT, and TRT. RRT is the time it takes for a participant to notice the light (i.e., the time between stimulus onset and the participant lifting his or her finger from the start button). MRT indexes the movement component of this task and is the time between the participant lifting his or her finger from the start button and touching the response button. TRT is the sum of RRT and MRT.
Mean TA_AUE of percentage correct response relative to CRT score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The CRT task is a classic test of reaction time used to measure psychomotor performance. During this test, the participant is presented with an onscreen equivalent of the numeric keypad. The participant must quickly press the buttons on a separate keypad that corresponds with the keys illuminated on the screen. The CRT task comprises 3 outcome variables: RRT, MRT, and TRT. RRT is the time it takes for a participant to notice the light (i.e., the time between stimulus onset and the participant lifting his or her finger from the start button). MRT indexes the movement component of this task and is the time between the participant lifting his or her finger from the start button and touching the response button. TRT is the sum of RRT and MRT.
CFBmax in Divided Attention (DA) score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The DA test is a manual-tracking test with a simultaneous visual target detection component. The participant is provided with a joystick with a trigger to execute this measure. During testing, the participant is presented with the image of an airplane and a randomly curving road. As the road moves down the screen, the participant is to try and position the image of the airplane over the center of the road.
Mean TA_AUE of DA score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The DA test is a manual-tracking test with a simultaneous visual target detection component. The participant is provided with a joystick with a trigger to execute this measure. During testing, the participant is presented with the image of an airplane and a randomly curving road. As the road moves down the screen, the participant is to try and position the image of the airplane over the center of the road.
CFBmin of percentage correct response relative to CRT score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The DA test is a manual-tracking test with a simultaneous visual target detection component. The participant is provided with a joystick with a trigger to execute this measure. During testing, the participant is presented with the image of an airplane and a randomly curving road. As the road moves down the screen, the participant is to try and position the image of the airplane over the center of the road.
Mean TA_AUE of percentage correct response relative to DA score (MRT subscale score, RRT subscale score, and TRT subscale score) | Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 (all Day 1), and 24 hours (Day 2) post-dose of each treatment cycle (up to 11 weeks)
  The DA test is a manual-tracking test with a simultaneous visual target detection component. The participant is provided with a joystick with a trigger to execute this measure. During testing, the participant is presented with the image of an airplane and a randomly curving road. As the road moves down the screen, the participant is to try and position the image of the airplane over the center of the road.
Number of participants with any treatment-emergent adverse event (TEAE) | Up to 20 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (Baseline) or: re-emerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment; or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants with any treatment-emergent serious adverse event (SAE) | up to 20 weeks
  A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (Baseline) or: re-emerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment; or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous. An SAE is any untoward medical occurrence that at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).

CONTACTS AND LOCATIONS:
Locations (1):
- INC Research Toronto, Inc., Toronto, Canada

REFERENCES:
- [Derived] Landry I, Hall N, Alur J, Filippov G, Reyderman L, Setnik B, Henningfield J, Moline M. Acute Cognitive Effects of the Dual Orexin Receptor Antagonist Lemborexant Compared With Suvorexant and Zolpidem in Recreational Sedative Users. J Clin Psychopharmacol. 2022 Jul-Aug 01;42(4):374-382. doi: 10.1097/JCP.0000000000001562. Epub 2022 Jun 24. PMID 35748777